CLINICAL TRIAL: NCT01252238
Title: Assessment of Renin Inhibition on Insulin Sensitivity, Diastolic Function and Aortic Compliance
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study sponsor terminated study due to AE's reported with valsartan and aliskiren
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Jonathan S. Williams, MD, MMSc, Jonathan Williams, MD, Brigham and Women's Hospital
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2010p001286
Record Dates: First submitted 2010-12-01; First posted 2010-12-02 (Estimated); Results first posted 2013-09-05 (Estimated); Last update posted 2018-02-13 (Actual); Status verified 2018-01

CONDITIONS: Insulin Sensitivity; Aortic Compliance; Diastolic Function
MeSH Terms: conditions — Insulin Resistance | interventions — aliskiren; Valsartan; Amlodipine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Valsartan and Aliskiren (Placebo Comparator): Valsartan 150 mg and Aliskiren (150 mg followed by force titration to 300 mg)
  Interventions: Drug: Valsartan and Aliskiren
- Aliskiren (Experimental)
  Interventions: Drug: Aliskiren
- Placebo Group (Placebo Comparator): Only taking Amlodipine
  Interventions: Drug: Amlodipine

INTERVENTIONS:
Drug: Aliskiren — Aliskiren 150 mg daily for 10 weeks, force titrated after initial 2 weeks.
  Arms: Aliskiren
Drug: Valsartan and Aliskiren — Subject taking combination of valsartan and aliskiren.
  Arms: Valsartan and Aliskiren
Drug: Amlodipine — Taking Amlodipine as prescribed by MD for management of high blood pressure.
  Arms: Placebo Group

SUMMARY:
This study is an investigation of the effect of commonly prescribed anti-hypertensive agents on insulin sensitivity, diastolic function and aortic compliance. The aims of the study are as follows:

Specific Aim 1: To determine in insulin resistant, hypertensive subjects if renin inhibition for 12 weeks modifies glucose homeostasis and insulin sensitivity.

To accomplish this specific aim, we will use three approaches: a fasting HOMA Index; and a three hour glucose tolerance test. Only hypertensive subjects with insulin resistance, as assessed by HOMA index will be enrolled in the study. Insulin resistance will be assessed basally and after twelve weeks of treatment with either a calcium channel blocker with placebo, or calcium channel blocker with a renin inhibitor, or a calcium channel blocker with a renin inhibitor and an angiotensin receptor antagonist.

Specific Aim 2: To determine in insulin resistant, hypertensive subjects if renin inhibition for 12 weeks modifies diastolic function and aortic compliance response to dietary sodium intake.

The same protocol and subjects will be used as defined in Specific Aim 1. Myocardial relaxation velocity (tissue Doppler imaging at the mitral annulus) and aortic compliance (characteristic aortic impedance) will be measured at baseline and then after acute and chronic renin inhibition:

1. Acute effect of renin inhibition: Hemodynamic measurements will be obtained on both high and low dietary sodium intake conditions (~1 week each) before and after a single dose of a renin inhibitor.
2. Chronic effect of renin inhibition: Hemodynamic measurements will be obtained at baseline and after 12 weeks of each of the three drug treatment arms above.

The study lasts 12 weeks and plans to study 45 hypertensive adults over the next two years.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, 18-70 years old
* BMI =/< 35
* BP: BP > 145/95 on no BP medication or on 3 or less BP medications
* HOMA =>2.5
* Any race

Exclusion Criteria:

* 4 or more BP medications
* Intolerance or known prior adverse history from taking the medications amlodipine, aliskiren or valsartan
* BP >170/110 on screening exam
* Alcohol intake >12 oz per week
* Current smoking
* Recreational drug use
* Known or suspected secondary hypertension
* Known history of coronary artery disease, cerebrovascular disease or congestive heart failure
* History or known kidney disease (eGFR <50cc/min)
* Diabetes or current metformin use, or HbA1c >=6.5% on screen
* Steroid use (oral or inhaled, chronic or within the past 6 months)
* Clinically significant screening lab abnormalities (See attached "Screening Labs Acceptable Ranges")
* Evidence of ischemia or heart block on screening electrocardiogram (greater than type I-second degree heart block, left bundle branch block, or ST-T wave changes in 2 or more contiguous leads).
* Acute hospitalizations including surgery in the past 6 months
* Chronic use of non-steroidal anti-inflammatory or narcotic medications
* Women who are pregnant or nursing, or wish to become pregnant and/or who can not agree or tolerate two forms of birth control during the study period:

Acceptable birth control methods for use in this study are:

* hormonal methods, such as birth control pills, patches, injections, vaginal ring, or implants
* barrier methods (such as a condom or diaphragm) used with a spermicide (a foam, cream, or gel that kills sperm)
* intrauterine device (IUD)
* abstinence (no sex)
* Significant concomitant medical illnesses (cancer, chronic active immunological conditions, etc.)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-06; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Williams, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred from 8/2009 thru 12/2011 at Brigham and Women's Hospital, Boston, MA.
Pre-assignment Details: All subjects washed out blood pressure medication for two weeks and ran in for two weeks on amlodipine 2.5-10mg titrated to BP <160/90 every other day. All subjects consumed a very low salt calculated diet for one week followed by calculated high salt diet for 2 weeks prior to randomization
Groups:
- Aliskiren: Aliskiren : Aliskiren 150 mg daily for 10 weeks, force titrated after initial 2 weeks.
- Placebo Group: Only taking Amlodipine
  Amlodipine : Taking Amlodipine as prescribed by MD for management of high blood pressure.
- Valsartan and Aliskiren: Valsartan 150 mg and Aliskiren (150 mg followed by force titration to 300 mg)
  Valsartan and Aliskiren : Subject taking combination of valsartan and aliskiren.
Period: Overall Study
Arm/Group | Aliskiren | Placebo Group | Valsartan and Aliskiren
Started | 8 | 8 | 8
Completed | 4 (sponsor terminated study) | 4 (sponsor terminated study) | 4 (sponsor terminated study)
Not Completed | 4 | 4 | 4
Not completed — Sponsor terminated study | 4 | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aliskiren | Placebo Group | Valsartan and Aliskiren | Total
Number analyzed (Participants) | 8 | 8 | 8 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 7 | 8 | 22
  >=65 years | 1 | 1 | 0 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (12) | 51 (6) | 47 (5) | 48 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 2 | 12
  Male | 4 | 2 | 6 | 12
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 8 | 24

OUTCOME MEASURES:

1. Primary Outcome: Change in Insulin Sensitivity by HOMA at 12 Weeks
Description: The difference (change) in HOMA calculated as Baseline HOMA minus 12-week HOMA value
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: HOMA Scale
Arm/Group | Aliskiren | Placebo Group | Valsartan and Aliskiren
Number analyzed (Participants) | 4 | 4 | 4
HOMA Scale | -0.7 (1.3) | -0.4 (1.4) | -0.5 (1.5)

2. Secondary Outcome: Aortic Compliance
Description: Characteristic aortic imedeance, dynes x s/cm5
Time Frame: 12 weeks
Population: Comparison of Baseline vs. study drug at 12 week2
Measure: Mean (Standard Error); unit: dyne x sec/cm5
Arm/Group | Valsartan and Aliskiren | Aliskiren | Placebo Group
Number analyzed (Participants) | 4 | 4 | 4
dyne x sec/cm5
  baseline | 212 (88) | 241 (63) | 111 (7)
  12 weeks | 174 (57) | 127 (0.00000) | 519 (499)

3. Other Pre Specified Outcome: Pulse Wave Velocity
Description: Measure of pulsewave velocity cm/s
Time Frame: 12 weeks
Population: Comparison of baseline vs at 12 weeks on study drug
Measure: Mean (Standard Error); unit: cm/s
Arm/Group | Valsartan and Aliskiren | Aliskiren | Placebo Group
Number analyzed (Participants) | 4 | 4 | 4
cm/s
  baseline | 991 (338) | 824 (106) | 1021 (5.6)
  12 weeks | 824 (183) | 696 (0.000000) | 574 (584)

ADVERSE EVENTS:
Arm/Group | Aliskiren | Placebo Group | Valsartan and Aliskiren
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8

LIMITATIONS AND CAVEATS:
No conclusions can be drawn from study due to very low sample size. The sponsor terminated the study after a separate study reported adverse events in a diabetic population who had taken both valsartan and aliskiren.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No